CLINICAL TRIAL: NCT02999568
Title: Open Study to Examine How Different Levels of Physical Activity Impact the Ovarian Reserve During the Pre-menopausal Period
Brief Title: The Effect of Exercise on Ovarian Reserve
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yael Pasternak, MD, Meir Medical Center
Other Study IDs: Meir Medical Center - Sport
Record Dates: First submitted 2016-12-15; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Physical Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: Women who practice high level of physical activity, as defined by International Physical Activity Questionnaire, for the past 3 years
  Interventions: Other: Physical exercise
- Control group: Women who practice low level of physical activity, as defined by International Physical Activity Questionnaire, for the past 3 years

INTERVENTIONS:
Other: Physical exercise — Women who practice high level of physical activity, as defined by International Physical Activity Questionnaire, for the past 3 years will be recruited. These women will will be asked to fulfill the International Physical Activity Questionnaire and additional questionnaire regarding relevant demographic and medical information. Blood samples to anti-mullerian hormone , leptin, and hormonal profile will be obtained in day 3 of menstruation. Ultrasound will be performed to measure Antral Follicular count and ovarian blood flow
  Groups: Experimental

SUMMARY:
The purpose of this study is to examine how different levels of physical activity impact the ovarian reserve during the pre-menopausal period

DETAILED DESCRIPTION:
Two groups are included:

1. The study group: women between 20-35 years of age who practice high level of physical activity, as defined by International Physical Activity Questionnaire , for the past 3 years
2. The control group: women between 20-35 years of age who practice low level of physical activity, as defined by International Physical Activity Questionnaire , for the past 3 years

Women who meet the criteria for inclusion for will be recruited to the study after signing a consent form. Recruitment will be done through sport centers. The control group will include women being examined in gynecologic emergency department, after signing a consent form, if they meet the control group's inclusion criteria. These women will be asked to fulfill the International Physical Activity Questionnaire and additional questionnaire regarding relevant demographic and medical information (see below). Blood samples to anti-mullerian hormone , leptin, and hormonal profile will be obtained in day 3 of menstruation. Ultrasound will be performed to measure Antral Follicular count and ovarian blood flow.

Data collection:

1. Demographic information on age, weight, height, BMI, marital status
2. Medical information regarding chronic diseases and medications
3. Obstetrical history
4. Information regarding physical activities in the version of International Physical Activity Questionnaire .
5. Information about menstrual behavior: irregularity (yes/no) frequency (less than 21 days between 21-35 days, over 35 days), menstrual duration (less than 3 days 3-7 days, or over 7 days) bleeding amount according to the number of pads per day (up to 1, 2, 4 or 5 pads).
6. Hormonal profile - Follicle-stimulating hormone , Luteinizing hormone , progesterone, Estradiol, Thyroid-stimulating hormone .
7. Antral Follicle Count, Anti-mullerian hormone
8. Leptin levels -reflecting metabolic changes.

ELIGIBILITY:
Inclusion Criteria:

Study group:

1. Women between 20-35 years of age who practice high level of physical activity, as defined by International Physical Activity Questionnaire, for the past 3 years
2. BMI 18-25
3. Regular menstruation

Control group:

1. Women between 20-35 years of age who practice low level of physical activity, as defined by International Physical Activity Questionnaire, for the past 3 years
2. BMI 18-25
3. Regular menstruation

Exclusion Criteria:

1. Polycystic ovary syndrome 2. Endometriosis 3. Diabetes 4. Hyper/hypothyroidism 5. BMI>25, BMI<18 6. Active or past eating disorder

-

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Control group - Recruitment will be done through Gynocologis tEmergency Experimental group - Recruitment will be done through sport centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-02; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Levels of anti-mullerian hormone | 3 days after period
Number of Antral Follicle Count | 3 days after period

SECONDARY OUTCOMES:
Levels of Follicle-stimulating hormone | 3 days after period
levels fo Luteinizing hormone | 3 days after period
Levels of progesterone | 3 days after period
Levels of estradiol | 3 days after period
Levels of Thyroid-stimulating hormone | 3 days after period
Levels of leptin | 3 days after period
Menstrual duration | 3 days after period
frequency of bleeding in every menstruation | 3 days after period
amount of bleeding in every menstruation | 3 days after period

CONTACTS AND LOCATIONS:
Overall Officials: Yael Pasternak, MD, Principal Investigator — Meir Medical Center

REFERENCES:
- [Background] Pate RR, Pratt M, Blair SN, Haskell WL, Macera CA, Bouchard C, Buchner D, Ettinger W, Heath GW, King AC, et al. Physical activity and public health. A recommendation from the Centers for Disease Control and Prevention and the American College of Sports Medicine. JAMA. 1995 Feb 1;273(5):402-7. doi: 10.1001/jama.273.5.402. PMID 7823386
- [Background] Clapp JF 3rd. Exercise during pregnancy. A clinical update. Clin Sports Med. 2000 Apr;19(2):273-86. doi: 10.1016/s0278-5919(05)70203-9. PMID 10740759
- [Background] Duckitt K. Exercise during pregnancy. BMJ. 2011 Sep 15;343:d5710. doi: 10.1136/bmj.d5710. No abstract available. PMID 21920880
- [Background] Rich-Edwards JW, Spiegelman D, Garland M, Hertzmark E, Hunter DJ, Colditz GA, Willett WC, Wand H, Manson JE. Physical activity, body mass index, and ovulatory disorder infertility. Epidemiology. 2002 Mar;13(2):184-90. doi: 10.1097/00001648-200203000-00013. PMID 11880759
- [Background] Oosthuyse T, Bosch AN. The effect of the menstrual cycle on exercise metabolism: implications for exercise performance in eumenorrhoeic women. Sports Med. 2010 Mar 1;40(3):207-27. doi: 10.2165/11317090-000000000-00000. PMID 20199120
- [Background] Clark AM, Ledger W, Galletly C, Tomlinson L, Blaney F, Wang X, Norman RJ. Weight loss results in significant improvement in pregnancy and ovulation rates in anovulatory obese women. Hum Reprod. 1995 Oct;10(10):2705-12. doi: 10.1093/oxfordjournals.humrep.a135772. PMID 8567797
- [Background] Hollmann M, Runnebaum B, Gerhard I. Effects of weight loss on the hormonal profile in obese, infertile women. Hum Reprod. 1996 Sep;11(9):1884-91. doi: 10.1093/oxfordjournals.humrep.a019512. PMID 8921059
- [Background] Morris SN, Missmer SA, Cramer DW, Powers RD, McShane PM, Hornstein MD. Effects of lifetime exercise on the outcome of in vitro fertilization. Obstet Gynecol. 2006 Oct;108(4):938-45. doi: 10.1097/01.AOG.0000235704.45652.0b. PMID 17012457
- [Background] Evenson KR, Calhoun KC, Herring AH, Pritchard D, Wen F, Steiner AZ. Association of physical activity in the past year and immediately after in vitro fertilization on pregnancy. Fertil Steril. 2014 Apr;101(4):1047-1054.e5. doi: 10.1016/j.fertnstert.2013.12.041. Epub 2014 Feb 10. PMID 24524834
- [Background] Masse LC, de Niet JE. Sources of validity evidence needed with self-report measures of physical activity. J Phys Act Health. 2012 Jan;9 Suppl 1:S44-55. doi: 10.1123/jpah.9.s1.s44. PMID 22287447